CLINICAL TRIAL: NCT05548881
Title: Implications of Maternal 45,X Mosaicism As A Secondary Genomic Finding Following Cell-free DNA Sequencing During Pregnancy: A Deep Phenotype Study
Status: Withdrawn | Type: Observational
Why Stopped: Study closed due to lack of resources. Study had no recruitment.
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000137; 000137-CH
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Phenotype; Metabolic Phenotype; Hypertensive Disease; Psychological Phenotype; Audio
Keywords: Fetal Neonatal; Maternal; Turner Syndrome; Chromosomes; reproductive; Natural History
MeSH Terms: conditions — Hypertension; Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Women who have submitted clinical samples for prenatal aneuploidy screening test with the finding of X mosaicism
- Group 2 (Control): Control group of Female volunteers of appropriate age, ethnicity, BMI, SES and parity

SUMMARY:
Background:

Mosaicism is a condition in which cells within the same person have a different genetic makeup. Sometimes, a type of mosaicism called 45,X may not be discovered in a woman until she undergoes routine tests during pregnancy. Little is known about how 45,X mosaicism may affect a person s long-term health.

Objective:

This natural history study will look for health risks in people with 45,X mosaicism.

Eligibility:

People aged 18 to 99 years who during pregnancy were found to have 45,X mosaicism. Healthy volunteers are also needed.

Design:

Participants will stay in the clinic for 2 days. They will have many tests:

A physical exam, including measurements of the body.

A gynecological exam, including genital measurements. Photos may be taken, with consent.

Blood tests, with blood drawn over an 8-week period. An oral glucose test for diabetes may also be done.

Tests of heart function. Participants will have small stickers attached to wires place on their chest, arms, and legs.

Hearing tests.

Ultrasound exams, which use echoing sound waves to create images of organs such as the heart and kidneys.

Imaging scans including x-rays, MRI, and DXA. The DXA uses x-rays to measure bone density and body fat. Other types of scans will capture images of the liver.

Participants will complete 4 surveys with questions about their sexual function, anxiety, depression, and health.

Participants may remain in the study for 20 years. For 5 years, they will have a yearly follow-up by phone or email. They may have follow-up visits at the clinic every 5 years.

DETAILED DESCRIPTION:
Study Description:

This is a deep phenotype study of women who are determined to have 45,X mosaicism as a secondary genomic finding following cfDNA sequencing during pregnancy.

Objectives:

* To define and describe a comprehensive phenotype of women with confirmed 45,X mosaicism initially found by cfDNA including cardiovascular, skeletal, metabolic, reproductive, audiometric, immunologic, and psychological functions.
* To compare the comprehensive phenotype of women with confirmed 45,X mosaicism with a control population (a. age and BMI-matched female controls without 45, X mosaicism at the initial visit and b. NHANES age-and BMI-matched female data for the applicable year.)
* To explore changes in phenotype for both 45,X mosaicism and control groups with somatic loss of X chromosome over time.

Endpoints:

Primary Endpoint: (i) Hypertension (as defined in 2017 by the American College of Cardiology/American Heart Association (ACC/AHA)

Secondary Endpoints:

* Cardiovascular:

  * Cardiac/coronary atherosclerosis
  * Cardiac function, valve assessment, aortic anatomy, endothelial function
* Skeletal:

  * Height
  * Areal bone mineral density (aBMD) as per DXA
  * Bone turnover markers
  * Bone microarchitecture using trabecular bone score as per DXA
  * Occult fractures using vertebral fracture assessment as per DXA
  * Skeletal morphology for assessment of scoliosis
* Metabolic:

  * Body fat distribution as per DXA
  * Anthropometrics; Body weight; Waist to hip ratio
  * Diabetes Mellitus
  * Thyroid disorders
  * Dyslipidemia
  * Assessment of liver for fatty disease and fibrosis as per abdominal MRE/MRS
* Gynecologic and urologic:

  * Markers of gonadal function and ovarian reserve
  * Primary ovarian insufficiency, Infertility, Early menopause as per participant history
  * Sexual function (as assessed by scores of the Female Sexual Function Index (FSFI) and the PROMIS(Registered Trademark) Sexual Function and Satisfaction Measures Version 2.0)
  * Ovarian and uterine imaging as per pelvic ultrasound.
  * Renal imaging as per renal ultrasound
* Obstetric:

  --Complications and outcomes of pregnancy as per participant history
* Audiometric:

  --Assessment of hearing loss
* Immunologic

  * Immune biomarkers
  * Celiac disease
* Psychological:

  * PROMIS(Registered Trademark) Item Bank v1.0 - Emotional Distress - Anxiety - Short Form 8a
  * PROMIS(Registered Trademark) Item Bank v.1.0 - Emotional Distress - Depression - Short Form 8b
  * PROMIS(Registered Trademark) Scale v.1.2 - Global Health

Exploratory endpoints: Changes in phenotype (as outlined above) for both 45,X mosaicism and control groups with somatic loss of X chromosome over time.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals of all races/ethnicities are eligible to participate.

* Individuals assigned female sex at birth ages >=18 to <= 99 years old who have not undergone medical and/or surgical transgender treatment
* Suspected maternal 45,X mosaicism as a secondary genomic finding following cfDNA sequencing during pregnancy
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Ability to read and comprehend written and verbal English as the documents required for the study have not been translated for non-English speaking speakers.

Inclusion criteria for control subjects:

* Individuals assigned female sex at birth ages >=18 to <= 99 years old who have not undergone medical and/or surgical transgender treatment
* Good general health. In general, subjects should take no medications. The use of over the counter and prescription medications will be reviewed on a case-by-case basis; depending on the medication, subjects who have continued to take prescription medication prior to study entry may be still eligible.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Ability to read and comprehend written and verbal English as the documents required for the study have not been translated for non-English speaking speakers.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria at screening or baseline will be excluded from participation in this study:

* Male and transfemale individuals
* Individuals with significant medical comorbidities (e.g. NYHA Class III or IV heart failure, or CKD Stage 3b or worse (eGFR < 60 mL/min/1.73 m2), or American Society of Anesthesiologists Physical Status Class 3 or above) or other serious disorders at the discretion of the investigators.
* Individuals who have current substance abuse or a DSM 5 Axis I psychiatric disorder or DSM Axis II Mental Retardation diagnosis that in the opinion of the investigators would impede competence, compliance, or participation in the study

Exclusion criteria for control subjects:

* Male and transfemale individuals
* Individuals with significant medical comorbidities (e.g. NYHA Class III or IV heart failure, or CKD Stage 3b or worse (eGFR < 60 mL/min/1.73 m2), or American Society of Anesthesiologists Physical Status Class 3 or above) or other serious disorders at the discretion of the investigators.
* For females of reproductive potential: use of oral contraceptive pills, contraceptive patch, contraceptive vaginal ring within the past 3 months; use of depo medroxyprogesterone within the past 6 months; use of the etonorgestrel contraceptive implant within the past 1 month.
* Individuals who are pregnant, planning to become pregnant, currently nursing an infant, or have irregular menses, defined as cycles less than 21 days or greater than 45 days in premenopausal women.
* Previous history of the following: malignancy, chemotherapy, radiation therapy, primary ovarian insufficiency, galactosemia.
* Individuals who have current substance abuse or a DSM 5 Axis I psychiatric disorder or DSM Axis II Mental Retardation diagnosis that in the opinion of the investigators would impede competence, compliance, or participation in the study.
* Current use of tobacco or nicotine (eg. Nicotine patch, e-cigarette) products.
* Individuals who have had prior ear surgery other than myringotomy, individuals with cochlear implants, individuals who require use of hearing aids.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who have submitted clinical samples for prenatal aneuploidy screening test with the finding of X mosaicism will be recruited from laboratories that offer cell-free DNA testing during pregnancy as well as nation-wide obstetricians and maternal-fetal-medicine specialists Potential participants are likely to be referred from specialists who care for them or will find the protocol through an internet search A control group of volunteers of appropriate age, ethnicity, BMI, SES and parity will be recruited using resources of the NIH Office of Patient Recruitment (OPR) and AlescoData and will be a matched to study participants.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Hypertension | 5 Years
  Evaluation of hypertension as defined in 2017 by the American College of Cardiology/American Heart Association (ACC/AHA): Normal blood pressure - Systolic <120 mmHg and diastolic <80 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Gomez-Lobo, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Protocol does not specify IDP plans.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000137-CH.html